CLINICAL TRIAL: NCT01398033
Title: Paclitaxel-Coated Versus Uncoated Balloon for Treatment of Below-the-Knee In-Stent-Restenosis
Acronym: BAIR
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped due to lack of patient inclusion
Sponsor: Herz-Zentrums Bad Krozingen (Other)
Collaborators: University Heart Center Freiburg - Bad Krozingen (Other)
Responsible Party: Principal Investigator, Aljoscha Rastan, MD, Herz-Zentrums Bad Krozingen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FW-014-1
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: In-stent Stenosis of Infrapopliteal Arteries
Keywords: infrapopliteal arteries; In-stent stenosis; long lesions; drug-coated balloon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug-coated balloon (Active Comparator): 1. pre-dilatation of the target lesion with a non-coated balloon.
  2. treatment of the target lesion with the paclitaxel-coated balloon
  Interventions: Device: paclitaxel-coated balloon
- non-coated balloon (Placebo Comparator): Treatment of the target lesion with plain balloon angioplasty.
  Interventions: Device: non-coated balloon

INTERVENTIONS:
Device: paclitaxel-coated balloon — Balloon is coated with paclitaxel in a concentration of 3µg/mm2.
  Arms: Drug-coated balloon
Device: non-coated balloon — percutaneous transluminal angioplasty with a non-coated balloon
  Arms: non-coated balloon

SUMMARY:
There is both a poor life expectancy and a poor prognosis of limb salvage in those patience with stenoses or occlusions of the lower limb. To date only a small number of these patients could be helped through medication or surgery. The indications for stent placement are poor primary results following percutaneous transluminal angioplasty or evidence of a flow-limiting dissection. The primary success rate after a stent placement is between 80% and 90%. One so far inconsistent discussed problem is the occurrence of in-stent restenosis which is expected in 20% to 78% of treated lesions, depending on the stent used. Using only percutaneous transluminal angioplasty for treatment of an in-stent restenosis, restenosis reoccurs in 70% to 80% of cases.

The aim of this study is to analyse the primary success and the long term results of angioplasty using the drug-coated balloon (paclitaxel) compared to an non-coated balloon in the treatment of in-stent restenosis of lower limb arteries.

DETAILED DESCRIPTION:
In this prospective, double-blind, randomised, multi-centre study the use of the already certified coated balloon and an uncoated balloon is evaluated in patients with in-stent restenoses/reocclusions of the lower limb artery. The whole lesion length should be covered by the balloon so that proximal and distal overlap of the lesion by a minimum of 5mm is assured. Based on the current literature the average restenoses rate of the lower limb arteries after percutaneous transluminal angioplasty of an in-stent restenosis is 70% after 6 months. Assuming the restenosis rate reduces to 30% after percutaneous transluminal angioplasty using a drug-coated balloon, with a significance level of Alpha=0.05 (bilateral) and a power Beta=0.8, the enrolment of 100 patients is required in order to show a significant difference between treatment groups, considering a dropout rate of 30%. The choice of treatment will be distributed in a randomised, double blind procedure.

The study duration per patient is 2 years. Clinical follow-up evaluations will take place after 3 and 6 months and after 1 and 2 years. After 3 month and 12 months an angiography of the target vessel will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50 years
* Signed declaration of consent
* Subject is willing and able to participate in all the planned evaluations of the study protocol
* Arterial occlusion disease stage 3 - 6 Rutherford-Becker
* Subject with an in-stent stenosis over 70% of the vascular lumen diameter of the tibioperoneal trunc and/or the posterior tibial artery and/or of the anterior tibial artery and/or peroneal artery. Here vascular segments, which are affected continuous (including stent), proximal or distal of the stent by a relevant (re)stenosis, are treated according to randomisation
* The length of the target lesion(s) should not exceed 290mm
* In total four drug-coated balloons are enough to treat a maximum of two lesions
* The target lesion's lumen diameter is between 2.0mm and 3.5mm
* Successful passage of the wire to the target lesion before randomisation

Exclusion Criteria:

* Coagulopathy
* Pregnancy
* Contraindications for antiplatelet or heparin
* Factors which exclude a follow up
* Life expectancy <12 months
* Known allergies to contrast agents and/or Clopidogrel and/or Aspirin
* >50% stenosis distal of the target lesion
* Visible thrombus in the target lesion
* Lytic therapy 72 hours before the planned intervention
* Aneurysm of the femoral or popliteal artery
* Intervention of focal lesions of the femoral or popliteal artery may be carried out before treatment of the target lesion in order to enhance the inflow in the lower limb

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
primary patency of target lesion assessed by quantitative angiography | 3 months after index procedure

SECONDARY OUTCOMES:
Secondary patency of the target lesion assessed by quantitative angiography | 12 months after index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Aljoscha Rastan, M.D., Principal Investigator — Herzzentrum Bad Krozingen
Locations (1):
- Herzzentrum Bad Krozingen, Bad Krozingen, Germany